CLINICAL TRIAL: NCT02907346
Title: A Reinforcement Approach to Increase Use of CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1603017504; 1DP3DK097705-01 (NIH)
Record Dates: First submitted 2016-07-25; First posted 2016-09-20 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reinforcement for wearing CGM (Experimental): The intervention will reinforce patients for wearing CGM and for uploading it and reviewing its data.
  Interventions: Behavioral: Reinforcement for wearing CGM

INTERVENTIONS:
Behavioral: Reinforcement for wearing CGM — The intervention will reinforce patients for wearing CGM and for uploading it and reviewing its data.
  Other Names: Reinforcement for CGM wear

SUMMARY:
The purpose of this pilot project is to evaluate the effectiveness of a behavioral economic intervention to increase use of continuous glucose monitors (CGM) in adolescents and young adults with T1D. This study will be done in conjunction with Nancy Petry, PhD and her research team at University of Connecticut School of Medicine (UConn Health). The intervention will reinforce patients for wearing CGM and for uploading it and reviewing its data. A 6-month pilot trial will be conducted with up to 20 patients receiving the intervention. The specific aims are:

DETAILED DESCRIPTION:
The purpose of this pilot project is to evaluate the effectiveness of a behavioral economic intervention to increase use of continuous glucose monitors (CGM) in adolescents and young adults with T1D. This study will be done in conjunction with Nancy Petry, PhD and her research team at University of Connecticut School of Medicine (UConn Health). The intervention will reinforce patients for wearing CGM and for uploading it and reviewing its data. A 6-month pilot trial will be conducted with up to 20 patients receiving the intervention. The specific aims are:

1. To estimate how well a reinforcement intervention increases usage of CGM. The proportion of days on which participants wear the CGM will be determined as well as the number of weeks during which CGM is worn at least 5 days. We will compare usage rates in the pilot trial to historical control data of patients initiating CGM.
2. To evaluate the association between CGM usage and A1c. We expect A1c will decrease over time in patients who receive the reinforcement intervention. Patients who continue using the CGM are expected to have greater decreases in A1c than patients who discontinue its usage.

Evaluations will be conducted at time of CGM initiation, and 6, 13, 19, 26, and 39 weeks after treatment initiation to assess effects of the intervention and estimate effect sizes.

In addition to the primary aims, secondary outcomes will also be evaluated. Continued use of CGM is expected to improve aspects of diabetes management and daily functioning. Predictors of continued CGM usage and improvements in A1c will also be evaluated.

Results from this pilot study will be instrumental for guiding a subsequent, larger and longer term randomized study for evaluating reinforcement interventions for improving uptake of CGM, other diabetes-related adherence behaviors, and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. age 13-26 years old;
2. diagnosis of type 1 diabetes (T1D) >12 months via ADA guidelines
3. average A1c >7.5% and <14% during the year before study entry, and most recent A1c >7.5% but <14%;
4. have ordered and received a CGM, but have not used a CGM >3 days a week on average during the past 6 months.
5. test blood glucose levels at least 2 times per day on average;
6. access to a computer with internet for uploading CGM data;
7. access to a cell phone to communicate with research staff;
8. English speaking, able to read at >5th grade level, and pass an informed consent quiz; and adequate knowledge of insulin dosing and dietary recommendations for managing T1D.

Exclusion Criteria:

1. have a major psychiatric or neurocognitive disorder (e.g., severe learning impairment) that would inhibit participation;
2. have a major visual impairment;
3. have a significant other medical condition that impacts diabetes management (e.g., rheumatoid arthritis, or other condition that requires steroid treatment);
4. plan to switch insulin delivery mode (injection to pump or vice versa) in the next 12 months, or have recently switched.
5. Fail to complete the baseline phase wearing the CGM.

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the Proportion of days participants wear the CGM | up to 39 weeks
  CGM data uploaded to a CGM tracking website (e.g., Dexcom CLARITY™, Carelink) will be used to calculate the change in the proportion of days when the patient wore the CGM. At the 6, 13, 19, 26 and 39 week study visits, data will be uploaded and exported into an Excel file to calculate the days.
Change in the number of weeks participants wear the CGM on at least 5 days | up to 39 weeks
  CGM data uploaded to a CGM tracking website (e.g., Dexcom CLARITY™, Carelink) will be used to calculate the change in the number of weeks when the CGM is worn at least 5 days. At the 6, 13, 19, 26 and 39 week study visits, CGM data will be uploaded and exported into an Excel file to calculate the number of weeks when it is worn at least 5 days.
Change in A1c | up to 39 weeks
  Change in A1c will be evaluated at the week 6, 13, 19, 26 and 39 week study visits by finger prick (DCA Vantage,Siemons).

CONTACTS AND LOCATIONS:
Overall Officials: William Tamborlane, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No